CLINICAL TRIAL: NCT02197624
Title: Metabolic Adaptation to Plant-based Diets in Asian Populations
Brief Title: Genetic Variants and Iron Absorption
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB #: 1206003117
Record Dates: First submitted 2014-07-16; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Iron Absorption
Keywords: Non-heme iron absorption; HFE

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two 10 mL blood samples and one 3 mL blood sample were collected.
Oversight: Data Monitoring Committee: No

SUMMARY:
The two specific aims of this study are: 1) to assess the impact of a genetic variant on iron status; 2) to assess the impact of a genetic variant on non-heme absorption among Asian women. The investigators hypothesize that the genetic variant could enhance iron status and iron absorption in Asian women.

DETAILED DESCRIPTION:
To determine the HFE genotype of female Asian study volunteers, we collected venous blood samples and extracted DNA from these blood samples. HFE genotype was determined as CC, CT, and TT and used to assess possible differences in iron status as a function of genotype. To measure the impact of genotype on non-heme Fe absorption, a sub-group of women with the CC (n=10) or TT (n=11) genotype were invited to return for an Fe absorption study. Each volunteer consumed stable 57Fe (as ferrous sulfate). Two weeks after ingesting this tracer, a blood sample was collected from each woman and the amount of non-heme (57Fe) iron incorporated into red blood cells was measured with magnetic sector thermal ionization mass spectrometry. Possible associations between iron status and iron absorption as a function of genotypes were explored. Data from this study will provide information that aims to improve human health by better understanding the iron requirements of individuals with different genetic background.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant and between the ages of 18~35 y
* East Asian descent with both maternal and paternal grandparents from East Asia, including China, Japan, South Korea, Vietnam, Thailand, Malaysia and Singapore

Exclusion Criteria:

* taking or planing to take any vitamin or mineral supplements during the study period
* pre-existing medical problems that might impact inflammation or Fe status, including malabsorption, blood disorders, ulcers, joint diseases and asthma
* taking any prescribed medications known to affect iron homeostasis

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women were eligible for the study if they met the following criteria: 1) non-pregnant and between the ages of 18~35 y; 2) of East Asian descent with both maternal and paternal grandparents from East Asia, including China, Japan, South Korea, Vietnam, Thailand, Malaysia and Singapore; 3) not taking any vitamin or mineral supplements for at least 1 month before the study and during the 2-week study interval; 4) no pre-existing medical problems including malabsorption, blood disorders, ulcers, joint diseases or asthma that might impact inflammation or Fe status; 5) not taking any prescribed medications known to affect iron homeostasis.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Genotype at SNP rs9366637 | 2 weeks after the participant's visit to the laboratory
  At the participant's visit to the laboratory, a 10 mL blood sample was collected. The blood sample was used for determining genotype.
Hemoglobin | Up to 2 days after the participant's visit to the laboratory
  At the participant's visit to the laboratory, a 10 mL blood sample was collected. The blood sample was used for determining the concentration of hemoglobin.
Serum Ferritin | Up to 6 months after the participant's visit to the laboratory
  At the participant's visit to the laboratory, a 10 mL blood sample was collected. The blood sample was used for determining the concentration of serum ferritin.
Serum transferrin receptor | Up to 6 months after the participant's visit to the laboratory
  At the participant's visit to the laboratory, a 10 mL blood sample was collected. The blood sample was used for determining the concentration of serum transferrin receptor.
Non-heme Iron absorption in women with 2 HFE genotypes | one month for screening with genotype then 2 weeks for iron absorption study
  Women donated a blood sample for genotyping. Women with particular HFE genotypes were invited to return for an absorption study. Two weeks after women consume the iron tracer, a blood sample was obtained to measure the amount of iron absorbed.

SECONDARY OUTCOMES:
Folate | Up to 6 months after the participant's visit to the laboratory
  At the participant's visit to the laboratory, a 10 mL blood sample was collected. The blood sample was used for determining the concentration of folate.
Vitamin B-12 | Up to 6 months after the participant's visit to the laboratory
  At the participant's visit to the laboratory, a 10 mL blood sample was collected. The blood sample was used for determining the concentration of vitamin B-12.
C-reactive protein | Up to 6 months after the participant's visit to the laboratory
  At the participant's visit to the laboratory, a 10 mL blood sample was collected. The blood sample was used for determining the concentration of C-reactive protein.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly O'Brien, PhD, Principal Investigator — Cornell University
Locations (1):
- Human Metabolic Research Unit, Cornell University, Ithaca, New York, United States